CLINICAL TRIAL: NCT07047235
Title: Understanding Substrate Evolution in Persistent Atrial Fibrillation to Develop Tailored Ablation Strategies
Brief Title: Substrate Remodelling and Targeted Ablation in AF
Acronym: STRATA-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 407
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation (AF); Atrial Fibrillation Mechanisms; Catheter Ablation; Low Voltage Areas
Keywords: ganglionic plexi; autonomic remodelling; substrate remodelling; conduction velocity
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This study is a single-centre, prospective mechanistic cohort investigation with a nested interventional controlled study designed to comprehensively evaluate electrophysiological substrate remodelling and its relationship with procedural outcomes in patients undergoing catheter ablation for persistent AF.
  Patients already undergoing a first ablation for persistent atrial fibrillation will undergo extensive structural, electrical and autonomic modelling during their index ablation procedure. They will then be followed up for 1 year.
  Those whose AF recurs will be invited for a repeat procedure in which all patients will undergo reisolation of the pulmonary veins and ganglionic plexi. Those whose atria is comprised of low voltage zones more than 30 will additionally undergo susbtrate modification of rate dependent conduction velocity slowing sites. All these patients will then undergo further follow up for 12 months will be compared to propensity matched controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimal Low Voltage Zones Group (Active Comparator): These are patients who've had recurrence of AF after their first ablation and less than 30% of their atria is comprised of low voltage zones. They will undergo autonomic ganglionic plexi site ablation combined with pulmonary vein re-isolation.
  Interventions: Procedure: Pulmonary vein reisolation; Procedure: Ganglionic plexi ablation
- Significant Low Voltage Zones Group (Active Comparator): These are patients who've had recurrence of AF after their first ablation and greater than 30% of their atria is comprised of low voltage zones. They will undergo targeted ablation of conduction slowing sites in addition to ganlionic plexi site ablation and pulmonary vein reisolation.
  Interventions: Procedure: Pulmonary vein reisolation; Procedure: Ganglionic plexi ablation; Procedure: Substrate ablation

INTERVENTIONS:
Procedure: Pulmonary vein reisolation — The pulmonary veins will be checked electrically and further ablation will be undertaken if they are not isolated.
Procedure: Ganglionic plexi ablation — Sites where ganglionix plexi have been found will be ablated.
Procedure: Substrate ablation — Areas of rate dependent conduction velocity slowing will be targeted using cathether ablation
  Arms: Significant Low Voltage Zones Group

SUMMARY:
Atrial fibrillation (AF) is the most common heart rhythm disorder, affecting millions worldwide and causing symptoms such as palpitations, fatigue and breathlessness. It also increases the risk of stroke and heart failure, so effective treatment is essential.

A treatment for AF involves catheter ablation, a minimally invasive procedure where problematic areas of the heart are targeted using controlled energy. This is done by passing wires called catheters, through blood vessels at the top of the leg all the way to the heart. However, this isn't effective for everyone and approximately half of patients experience a return of AF despite treatment.

In this researcher-led study at St Bartholomew's Hospital , the investigators will use a method called electroanatomical mapping to make a 3D picture of the left atrium, the heart's upper left chamber. To make this picture more detailed, information will be collected - such as how strong electrical signals are (voltage), how fast and in which direction they travel through the heart to describe abnormal areas and areas of scar within the heart. Information will also be gathered about the routes electricity takes and the nerve activity in the heart muscle. These detailed maps will help to understand why AF can continue indefinitely in some people, why ablation works for some people and not others, and improve how ablations are done to make them more effective.

All participants will undergo catheter ablation with these mapping methods integrated into the procedure. If AF recurs, patients will be invited for a second ablation targeting specific abnormal areas depending on the amount of scar found. This will be standardised across patients.

Patients will be followed for 12 months, with structured visits at 3, 6, 9 and 12 months and 48-hour ECG recorders at 6 and 12 months. By tracking how the heart's structure and electrical behaviour evolve, the aim is to to see if map-guided ablation reduces the need for further procedures, lowers healthcare costs and improves quality of life.

Ultimately, this study will provide clear, reproducible insights into AF mechanisms and yield practical guidance so clinicians can predict who will benefit from standard ablation treatment and who may require extra, map-guided treatment.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent
* Age: 18 years or older
* Clinical diagnosis: Persistent atrial fibrillation
* Treatment status: Scheduled to undergo first-time catheter ablation for persistent AF

Exclusion Criteria:

* Inability or unwillingness to provide informed consent
* Under 18 years of age
* Previous left atrial ablation for AF or other atrial arrhythmias
* Any clinical contraindications to undergoing AF catheter ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2029-11-18 (Estimated); Study Completion 2030-08-18 (Estimated)

PRIMARY OUTCOMES:
Assessment of Electrical, Structural and Autonomic Remodelling in Persistent Atrial Fibrillation | 4 years
  A primary objective of this study is to delineate the remodelling changes that occur in persistent atrial fibrillation and to utilise these to develop tailored ablation strategies.
Establish a Predictive Model to Idenitfy Which Patients are Responders to Pulmonary Vein Isolation Alone and Who Will Require Further Tailored Ablation Strategies | 24 months
  Based on clinical data approximately only 50% of patients with persistent atrial fibrillation who undergo pulmonary vein isolation remain in sinus rhythm. A main aim of the study is to develop a method to identify which patients will respond to pulmonary vein isolation alone and who will require further tailored ablation strategies.
To Assess if Ablation of Rate Dependent Conduction Velocity Slowing Sites Improves Freedom from Atrial Fibrillation | 5 years
  All patients who recur after their initial ablation will be invited to undergo a repeat ablation procedure. All patients will undergo ganglionic plexi ablation and reisolation their pulmonary veins. Those who have low voltage zones of more than 30% of their total left atrium will undergo further ablation of rate dependent conduction velocity slowing sites.

SECONDARY OUTCOMES:
Develop Personalised Electrical Atrial Models | 5 years
  The data taken from the electrophysiological procedures will be used to create mathematical computer models that can be used as an environment to test electrophysiological theories and response to ablation.

CONTACTS AND LOCATIONS:
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No